CLINICAL TRIAL: NCT00988715
Title: Hematopoietic Cell Transplantation for Patients With High-Risk Acute Myeloid Leukemia (AML), Acute Lymphoblastic Leukemia (ALL), or Myelodysplastic Syndrome (MDS) Using Radiolabeled DOTA-Biotin Pretargeted by BC8 Antibody-Streptavidin Conjugate
Brief Title: Donor Peripheral Blood Stem Cell Transplant and Pretargeted Radioimmunotherapy in Treating Patients With High-Risk Advanced Acute Myeloid Leukemia, Acute Lymphoblastic Leukemia, or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2309.00; NCI-2009-01294 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2309.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P01CA044991 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Chronic Myelomonocytic Leukemia; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Previously Treated Myelodysplastic Syndrome; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Refractory Anemia With Excess Blasts; Refractory Cytopenia With Multilineage Dysplasia; Refractory Cytopenia With Multilineage Dysplasia and Ringed Sideroblasts; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Myeloproliferative Disorders; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts | interventions — Cyclosporine; Cyclosporins; Mycophenolic Acid; Whole-Body Irradiation; Peripheral Blood Stem Cell Transplantation; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (PRIT, transplant) (Experimental): Patients undergo pretargeted radioimmunotherapy comprising a test dose of BC8-SA conjugate IV on day -22 and 111In-DOTA-biotin IV on day -20, followed by a therapy dose of BC8-SA conjugate IV on day -14 and 90Y-DOTA-biotin IV on day -12. Patients receive fludarabine phosphate IV on days -4 to -2. Patients undergo TBI and then peripheral blood stem cell transplant on day 0. Patients with matched related donors receive cyclosporine IV on days -3 to 56 and taper to day 180 and mycophenolate mofetil PO BID on days 0-27. Patients with matched unrelated donors receive cyclosporine IV on days -3 to 100 and taper to day 180 and mycophenolate mofetil PO TID on days 0-40 and taper to day 96.
  Interventions: Biological: Pretargeted Radioimmunotherapy; Drug: Cyclosporine; Drug: Mycophenolate Mofetil; Radiation: Total-Body Irradiation; Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Fludarabine Phosphate; Other: Pharmacological Study; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Pretargeted Radioimmunotherapy — Antibody-streptavidin conjugate and radiolabeled DOTA-biotin, each given IV
Drug: Cyclosporine — Given IV
  Other Names: 27-400; CsA; Neoral; OL 27-400; Sandimmun
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
Radiation: Total-Body Irradiation — Undergo total-body irradiation
  Other Names: TBI; Total Body Irradiation; Whole-Body Irradiation
Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation — Undergo peripheral blood stem cell transplant
  Other Names: Non-myeloablative allogeneic transplant; Nonmyeloablative Stem Cell Transplantation; NST
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo peripheral blood stem cell transplant
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; SH T 586
Other: Pharmacological Study — Correlative studies
  Other Names: pharmacological studies
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial studies pretargeted radioimmunotherapy and donor peripheral blood stem cell transplant employing fludarabine phosphate and total-body irradiation (TBI) to treat patients with high-risk acute myeloid leukemia, acute lymphoblastic leukemia, or myelodysplastic syndrome. Giving chemotherapy drugs, such as fludarabine phosphate, and TBI before a donor peripheral blood stem cell transplant helps stop the patient's immune system from rejecting the donor's stem cells. Radiolabeled monoclonal antibodies can be combined with fludarabine phosphate and TBI to find cancer cells and kill them without harming normal cells. Pretargeted radioimmunotherapy (PRIT) allows for further improved targeting of tumor cells over standard directly labeled antibodies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) of radiation delivered via PRIT using BC8-SA (BC8 antibody-streptavidin conjugate) when combined with fludarabine (FLU) (fludarabine phosphate), 2 Gy total body irradiation (TBI), cyclosporine (CSP), mycophenolate mofetil (MMF), and allogeneic hematopoietic cell transplant (HCT) in patients who have advanced acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), or high risk myelodysplastic syndromes (MDS).

SECONDARY OBJECTIVES:

I. To estimate rates of immune reconstitution, engraftment, and donor chimerism resulting from this combined preparative regimen.

II. To estimate rates of disease relapse, acute graft-versus-host disease (GvHD), and day-100 disease-free survival in patients receiving PRIT using BC8-SA combined with FLU, 2 Gy TBI, CSP, MMF, and allogeneic HCT.

III. To assess biodistribution, serum half-life, urinary excretion, tissue localization, and clearance of BC8-SA conjugate and DOTA-biotin.

IV. To assess the feasibility of yttrium y 90 (90Y)-DOTA-biotin to bind to BC8-SA conjugate localized to hematolymphoid tissues.

OUTLINE:

Patients undergo pretargeted radioimmunotherapy comprising a test dose of BC8-SA conjugate intravenously (IV) on day -22 and indium In 111(111In)-DOTA-biotin IV on day -20, followed by a therapy dose of BC8-SA conjugate IV on day -14 and 90Y-DOTA-biotin IV on day -12. Patients receive fludarabine phosphate IV on days -4 to -2. Patients undergo TBI and then peripheral blood stem cell transplantation on day 0. Patients with matched related donors receive cyclosporine IV on days -3 to 56 and taper to day 180 and mycophenolate mofetil orally (PO) twice daily (BID) on days 0-27. Patients with matched unrelated donors receive cyclosporine IV on days -3 to 100 and taper to day 180 and mycophenolate mofetil PO thrice daily (TID) on days 0-40 and taper to day 96.

After completion of study treatment, patients are followed up at 6, 9, 12, 18, and 24 months, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced AML or ALL defined as beyond first remission, primary refractory disease, or evolved from myelodysplastic or myeloproliferative syndromes; or patients with MDS expressed as refractory anemia with excess blasts (RAEB), refractory cytopenia with multilineage dysplasia (RCMD), RCMD with ringed sideroblasts (RCMD-RS), or chronic myelomonocytic leukemia (CMML)
* Patients not in remission must have CD45-expressing leukemic blasts; patients in remission do not require phenotyping and may have leukemia previously documented to be CD45 negative (because in remission patients, virtually all antibody binding is to nonmalignant cells which make up >= 95% of nucleated cells in the marrow)
* Patients should have a circulating blast count of less than 10,000/mm^3 (control with hydroxyurea or similar agent is allowed)
* Patients must have an estimated creatinine clearance greater than 50/mL per minute
* Bilirubin < 2 times the upper limit of normal
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2 times the upper limit of normal
* Karnofsky score >= 70 or Eastern Cooperative Oncology Group (ECOG) =< 2
* Patients must have an expected survival of > 60 days and must be free of active infection
* Patients must have an human leukocyte antigen (HLA)-identical sibling donor or an HLA-matched unrelated donor who meets standard Seattle Cancer Care Alliance (SCCA) and/or National Marrow Donor Program (NMDP) or other donor center criteria for peripheral blood stem cell (PBSC) donation; related donors should be matched by molecular methods at the intermediate resolution level at HLA-A, B, C, and DRB1 according to Fred Hutchinson Cancer Research Center (FHCRC) Standard Practice Guidelines and to the allele level at DQB1; unrelated donors should be identified using matching criteria that follows the FHCRC standard practice guidelines limiting the study to eligible donors that are allele matched for HLA-A, B, C, DRB1, and DQB1 (Grade 1), and accepting up to one allele mismatch as per standard practice grade 2.1 for HLA-A, B, or C; PBSC is the only permitted stem cell source
* DONOR: Donors must meet HLA matching criteria as well as standard SCCA and/or NMDP, or other donor center criteria for PBSC donation

Exclusion Criteria:

* Circulating human anti-mouse antibody (HAMA) or human anti-streptavidin antibody (HASA)
* Prior radiation to maximally tolerated levels to any critical normal organ
* Patients may not have symptomatic coronary artery disease and may not be on cardiac medications for anti-arrhythmic or inotropic effects
* Patients with the following organ dysfunction:

  * Left ventricular ejection fraction < 35%
  * Corrected diffusion capacity of the lung for carbon monoxide (DLCO) < 35% and/or receiving supplemental continuous oxygen
  * Liver abnormalities: fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction as evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis, or symptomatic biliary disease
* Patients who are known seropositive for human immunodeficiency virus (HIV)
* Perceived inability to tolerate diagnostic or therapeutic procedures, particularly treatment in radiation isolation
* Active central nervous system (CNS) leukemia
* Women of childbearing potential who are pregnant (beta-human chorionic gonadotropin [b-HCG] +) or breast feeding
* Fertile men and women unwilling to use contraceptives during and for 12 months post-transplant
* Patients may not use vitamin supplements containing biotin from the time of 1 week prior to treatment until 1 week after completion of treatment with all PRIT components
* Inability to understand or give an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-04-21 (Actual); Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLT) (grade III/IV Bearman) to determine MTD of radiation delivered to normal organ by pretargeted 90Y-DOTA-biotin | Within 100 days post-transplant
  Conducted by the "two-stage" approach introduced by Storer. The MTD will be defined as the dose of 90Y-DOTA-biotin used in combination with the non-myeloablative HCT conditioning regimen that is associated with a grade III/IV regimen related toxicity (RRT) or true DLT rate of 25%.

SECONDARY OUTCOMES:
Rates of engraftment, chimerism, and non-relapse mortality | Days 28
  Chimerism testing methods will be in accordance with Standard Practice Guidelines, with timing consistent with other non-myeloablative transplant protocols. Mixed or full donor chimerism will be evidence of donor engraftment. Full Chimerism is defined as > 95% donor CD3+ T cells and mixed chimerism is the detection of peripheral blood donor T cells (CD3+) and granulocytes (CD33+) as a proportion of the total peripheral blood T cell and granulocyte population, respectively. The true rate of graft rejection exceeds must be less than 20%.
Rates of engraftment, chimerism, and non-relapse mortality | Day 84
  Chimerism testing methods will be in accordance with Standard Practice Guidelines, with timing consistent with other non-myeloablative transplant protocols. Mixed or full donor chimerism will be evidence of donor engraftment. Full Chimerism is defined as > 95% donor CD3+ T cells and mixed chimerism is the detection of peripheral blood donor T cells (CD3+) and granulocytes (CD33+) as a proportion of the total peripheral blood T cell and granulocyte population, respectively. The true rate of graft rejection exceeds must be less than 20%.
Rate of grades III-IV acute GVHD | At day +100
  Graded according to the established criteria at the FHCRC.
Achievement and duration of response | Up to 24 months
  Complete remission is defined as complete resolution of all signs of myelodysplasia or leukemia for at least four weeks with normal bone marrow with blasts < 5% with normal cellularity, normal megakaryopoiesis, more than 15% erythropoiesis, and more than 25% granulocytopoiesis; normalization of blood counts; and no extramedullary disease. Partial remission is defined as improvement of hematological parameters in the peripheral blood and 50% decline in marrow blasts from pre-transplant level with > 10% erythropoiesis and 25% granulocytopoiesis.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Sandmaier, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States